CLINICAL TRIAL: NCT04620421
Title: Effect of Rhythm-based Multitask Training on Fall Rate in Community-dwelling Older Adults: An Assessor-blinded, Randomized, Controlled Trial
Brief Title: Effect of Rhythm-based Multitask Training on Falls Among Older Adults
Acronym: RYMA
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Jens Eg Nørgaard, PhD-student, Cand.Scient., Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N-20200019
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Accidental Fall; Fall Injury
Keywords: Older adults; Dual-task; Gait adaptability; Multitask; Music-based exercise; Fall prevention; Exercise; Quality of Life; Dalcroze Eurhythmics
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: After baseline assessments, participants will be randomly allocated to either the training or control group. To produce groups of similar size a permuted block randomization will be used. Allocation concealment will be maintained using random block sizes (4, 6, or 8) and by the randomization code only being available for non-blinded research staff.
  The intervention group will undergo 6 months of RYMA training, meanwhile, the control group will continue their regular activity schedule.
Who Masked: Outcomes Assessor
Masking Description: The randomization will be conducted by staff members not involved in the data collection. Moreover, the randomization code will only be available for non-blinded research staff to maintain allocation concealment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Rhythm-based multitask training) (Experimental): Randomized to participate in the rhythm-based multitask training intervention
  Interventions: Other: Rhythm-based Multitask Training
- Control group (Continuation of regular activity schedule) (No Intervention): Randomized to the control group who is encouraged to continue their regular everyday routines, which may include self-administrated training exercises.

INTERVENTIONS:
Other: Rhythm-based Multitask Training — Participants will be assigned to a weekly one-hour RYMA session for six months, followed by a six-month follow-up period without training. An experienced instructor will perform the RYMA sessions, which consists of a wide variety of rhythm-based multitask exercises performed to improvised piano music. The RYMA intervention is inspired by Dalcroze eurhythmics and exercises consists of components such as 1) coordination between hands and/or feet, 2) dissociation between hands and/or feet, 3) movements based on musical cues (e.g. follow the tempo), 4) movement inhibition based on musical cues, 5) handling of props (e.g. balls, scarfs, and plates), 6) pair or group-based coordination movements (e.g. clapping each other's hands and mirroring movements), 7) memorizing and repeating of rhythmic patterns, and 8) quick motoric responses to unexpected cues.
  Arms: Training group (Rhythm-based multitask training)

SUMMARY:
In this assessor-blinded, randomized, controlled trial our primary aim is to quantify the effects of a six-month rhythm-based multitask training (RYMA) intervention on fall rates collected over 12 months, compared to continuation of regular activity schedule, among community-dwelling older adults (≥70 years).

This assessor-blinded, randomized, controlled trial aim is to quantify the effects of six-month rhythm-based multitask training (RYMA) on fall rates collected over 12 months, compared to continuation of regular activity schedule, among community-dwelling older adults (≥70 years).

A sample size calculation estimates that 126 older community-dwelling older adults (≥70 years) are needed. Following baseline measures, the recruited participants will randomly be assigned to either the RYMA or the control group. The participants in the RYMA group will be assigned to a single weekly one-hour session for six months, while the control group will be encouraged to continue their regular activity schedule. Assessment of the primary outcome, fall rates, will be conducted continuously in 12 months from the beginning of training using monthly fall calendars. When a fall is reported in the fall calendar, a telephone interview will be conducted to assess circumstances and consequences (e.g. fall-related fractures, fall-related hospital admissions) of the falls. Moreover, assessment of physical, cognitive, and social-psychological surrogate outcomes will be made at baseline, six, and 12 months.

DETAILED DESCRIPTION:
Background:

Approximately one-third of older adults (≥65 years) fall at least once a year and 40-60% of falls lead to injuries. Of these injuries, 30-40% are minor, such as brushes, while 10% are serious, such as head injuries or fractures. Indeed, falls are the most common cause of injuries among older adults, and injuries are the fifth leading cause of premature death among older adults.

In an attempt to reduce the fall rate, several fall prevention interventions have been examined. Here, physical exercise has proven as an effective and cost-effective approach. However, the majority of exercise interventions only addressed physical risk factors while only a few focused on cognitive risk factors. For instance, a reduced executive function has been associated with increased fall risk. Thus, interventions addressing both physical and cognitive functions could enhance the efficacy of fall prevention.

Cognitive-motor training is a training modality that simultaneously incorporates physical and cognitive elements. A cognitive-motor training approach is RhYthm-based Multitask trAining (RYMA). During RYMA, participants perform rhythm-based balance-challenging multitask exercises following the rhythm of improvised piano music. A preliminary study by Trombetti et al. 2011 showed promising results as the fall rate decreased by 54% following six months of RYMA using a Dalcroze Eurhythmics approach compared to controls. The observed reduced fall rate may be due to RYMAs ability to decrease gait variability under dual-task conditions, improve postural balance, and executive function. However, the Trombetti study had some limitations. For instance, the primary outcome was gait-variability and not fall rates. Thus, the study was not adequately designed to quantify differences in fall rates (e.g. no follow-up period with a no-attention control group). Moreover, the effects of RYMA on social-psychological factors, such as health-related quality of life (HRQoL), fear of falling, and loneliness is yet be investigated.

Methods:

This assessor-blinded, randomized, controlled trial primarily aims to quantify the effects of a six-month RYMA intervention on fall rates collected over 12 months compared to continuation of regular activity schedule, among community-dwelling older adults (≥70 years). Secondly, we want to evaluate the effects of RYMA on fall risk, fall-related fractures, fall-related hospital admissions, as well as physical, cognitive, and social-psychological factors to explain potential mechanisms concerning fall rate.

Community-dwelling older adults, the municipality of Aalborg will be recruited through appetizers of RYMA, flyers, and advertisements in local newspapers, radio, and television. After baseline assessments, participants will be randomly allocated to either the RYMA or control group. The participants in the RYMA group will be assigned to a single weekly one-hour session for six months, while the control group will be encouraged to continue their regular activity schedule., which may include self-administrated training exercises. The primary outcome, fall rate (falls per person-year), will be assessed continuously from the day of the baseline assessments and for 12 months after the RYMA intervention begins using monthly fall calendars in line with the recommendation. In the present study, a fall will be defined as "an unexpected event in which the participant comes to rest on the ground, floor, or lower-level". When a fall is reported in the fall calendar, a telephone interview will be conducted to assess circumstances and consequences (e.g. fall-related fractures, fall-related hospital admissions) of the falls. The secondary surrogate outcomes will be assessed at baseline, six, and 12 months. All data will be analyzed using an intention-to-treat approach.

A pilot study will be performed before the commencement of the study to evaluate the feasibility of employing RYMA at the senior activity centres and the acceptance of RYMA and the testing battery among participants. Thus, changes the protocol may be conducted based on the pilot study findings.

ELIGIBILITY:
Inclusion Criteria:

* ≥70 years old
* Community-dwelling
* Able to walk 20 meters without a walking aid
* Understand and remember a message in Danish
* Willing to provide informed consent for the trial

Exclusion Criteria:

* Having a progressive neurological disease (e.g. Parkinson, multiple sclerosis, etc.)
* Unstable medical conditions that would prevent safe participation
* Severe cognitive impairment
* Current participation in another fall prevention trial

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Fall rate (falls per person-years) | 12 months following the randomization
  Fall calendar

SECONDARY OUTCOMES:
Number of falls, number of fallers/non-/multiple-fallers, and time to first fall | 12 months following the randomization
  Fall calendar
Number of fall-related injuries | 12 months following the randomization
  Fall-calendar, verified by radiologically evidence
Number of fall-related hospital admissions | 12 months following the randomization
  Fall-calendar, verified by medical journals
Single- and dual-task gait | Baseline, six months, and 12 months
  8-meter gait test; dual-task: Serial subtractions by 3 from an random three-digit number
Single- and dual-task balance | Baseline, six months, and 12 months
  30-second static balance; dual-task: Grocery verbal fluency
Choice stepping reaction time | Baseline, six months, and 12 months
  Choice stepping reactions test on a Wii balance board
Lower extremity physical performance | Baseline, six months, and 12 months
  The Short Physical Performance Battery
Health-related quality of life | Baseline, six months, 12 months, and during phone-interview following a registered fall
  The EuroQoL EQ-5D-5L, Danish version
Fear of Falling | Baseline, six months, and 12 months
  The Short Falls Efficacy Scale international, Danish version
Loneliness | Baseline, six months, and 12 months
  The UCLA Loneliness Scale, Danish version
Executive function | Baseline, six months, and 12 months
  The Trail Making task Part A and B
Frailty | Baseline and 12 months
  The Tilburg Frailty Indicator

CONTACTS AND LOCATIONS:
Overall Officials: Jens E Nørgaard, Cand.Scient., Principal Investigator — Aalborg University Hospital
Locations (1):
- Department of Geriatric Medicine at Aalborg University, Aalborg, Northern Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No